CLINICAL TRIAL: NCT01090570
Title: Safety, Pharmacokinetic (PK), Pharmcodynamic (PD), and Drug-Drug Interaction of PLX3397 in Patients With Rheumatoid Arthritis Who Are Receiving Methotrexate
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Plexxikon (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PLX108-02
Record Dates: First submitted 2010-03-15; First posted 2010-03-22 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — pexidartinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- PLX3397 25 mg (Experimental)
  Interventions: Drug: PLX3397
- PLX3397 50 mg (Experimental)
  Interventions: Drug: PLX3397
- PLX3397 100 mg (Experimental)
  Interventions: Drug: PLX3397
- PLX3397 200 mg (Experimental)
  Interventions: Drug: PLX3397
- PLX3397 300 mg (Experimental)
  Interventions: Drug: PLX3397
- Placebo (Placebo Comparator)
  Interventions: Drug: PLX3397

INTERVENTIONS:
Drug: PLX3397 — Once-daily oral capsules

SUMMARY:
PLX3397 is a selective inhibitor of Fms and Kit activity. The objective of this study is to evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD), and drug-drug interaction (DDI) of orally administered PLX3397 during 2 weeks of dosing in patients with rheumatoid arthritis (RA) who are on maintenance methotrexate. This study is planned to provide data to inform dose selection for a subsequent 12 week dose ranging study in RA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years old with a diagnosis of rheumatoid arthritis by ACR criteria for ≥ 3 months.
* Prior to Baseline, patients must be on oral or subcutaneous methotrexate (≥ 10 mg/week and ≤ 25 mg/week) for at least 12 weeks (with a stable dose for at least 4 weeks) and folate (≥ 5 mg/week) for at least 6 weeks, and willing to continue on this regimen for the duration of the study.
* Adequate hematologic, hepatic, and renal function (absolute neutrophil count ≥ 1.5 X 109/L, Hgb > 9 g/dL, platelet count ≥ 100 X 109/L, AST/ALT WNL, albumin ≥ 3 g/dL, calculated CrCl>60 mL/min using Cockcroft-Gault formula).
* Women of child-bearing potential must have a negative pregnancy test within 7 days prior to initiation of dosing and must agree to use a double barrier method of birth control from the time of the negative pregnancy test up to 30 days after the last dose of study drug. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥1 year.
* Fertile men must agree to use an acceptable method of birth control while on study drug. Acceptable methods of contraception must include either abstinence from the first dose of study drug through 4 weeks after the last dose of study drug, or use of a condom with instructions to the female partner of child-bearing potential to also be protected as above.
* Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements.

Exclusion Criteria:

* Use of biologic response modifiers within the following periods prior to Day 1 Baseline: 4 weeks for Kineret (anakinra) and Enbrel (etanercept); 12 weeks for Remicade (infliximab), Humira (adalimumab), Simponi (golimumab), Orencia (abatacept), Actemra (tocilizumab), or Cimzia (certolizumab); 12 months for Rituxan.
* Use of Arava (leflunomide) within 12 weeks prior to Day 1 Baseline or any immunosuppressive agents other then hydroxychloroquine or sulfasalazine within 4 weeks of Day 1 Baseline.
* Investigational drug use within 4 weeks of Day 1 Baseline.
* Concomitant use of DMARDs (other than methotrexate), biological response modifiers, or known strong inducers or inhibitors of CYP3A4.
* Positive HepBsAg or HCV, or presence of clinically significant hepatic or biliary disease.
* Uncontrolled intercurrent illness.
* Refractory nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption.
* QTc ≥ 450 msec at Screening.
* The presence of a medical or psychiatric condition that, in the opinion of the Principal Investigator, makes the patient inappropriate for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To assess the drug-drug interaction of PLX3397 and Methotrexate in patients with rheumatoid arthritis | 2 weeks + 2 weeks follow up
  Blood samples will be taken at multiple time points during the 2 week time frame plus a 2 week follow up time frame to study the pharmacokinetics of PLX3397 and Methotrexate in patients.

SECONDARY OUTCOMES:
To assess the safety and tolerability of PLX3397 when taken once daily with concomitant methotrexate administration | 4 weeks
  Adverse events and safety lab tests (including a hematology panel, blood chemistry panel, coagulation and urinalysis) will be monitored throughout the study time frame.
To assess the pharmacokinetics of PLX3397 when taken once daily for 2 weeks at either a 25, 50, 100, 200 or 300 mg dose. | 2 weeks
  The pharmacokinetic profile of plasma PLX3397 will be analyzed by measurement of area under the plasma concentration-time curve (AUC0-t, AUC0-inf), peak concentration (Cmax), time to peak concentration (Tmax), half-life (t1/2), and terminal elimination rate constant (Kel).
To assess the pharmacodynamics of PLX3397 when taken once daily for 2 weeks at either a 25, 50, 100, 200 or 300 mg dose. | 4 weeks
  Measured by looking at the factors in the blood that may include, but are not limited to pro- and anti-inflammatory cytokines and mediators of the inflammatory process that may correlate with the activity of the disease and the response to PLX3397 in combination with methotrexate

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Tuscaloosa, Alabama
  - Little Rock, Arkansas
  - San Francisco, California
  - Altoona, Pennsylvania
  - Dallas, Texas